CLINICAL TRIAL: NCT01353001
Title: The Effect of Weight Loss and Exercise on Cardiovascular Disease Risk Factors in Class II and III Obese Women
Brief Title: Effect of Weight Loss on Cardiovascular Disease Risk Factors in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BSD-UPitt
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Cardiovascular Diseases
Keywords: Intervention Studies; Magnetic Resonance Imaging; C-Reactive Protein
MeSH Terms: conditions — Obesity; Cardiovascular Diseases | interventions — Diet; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diet Only (Experimental)
  Interventions: Behavioral: Diet
- Diet plus Aerobic Training (Experimental)
  Interventions: Behavioral: Diet Plus Aerobic Training
- Diet plus Resistance Training (Experimental)
  Interventions: Behavioral: Diet plus Resistance Training

INTERVENTIONS:
Behavioral: Diet — Participants will be given a calorie and fat gram goal according to their initial bodyweight. The fat gram goals will be set at 20% to 30% of total caloric intake. Subject calorie and fat gram goals are as follows: Subjects weighing less than 175 pounds will receive a diet prescription of 1200 calories and 27 fat grams per day. Subjects weighing between 175 and 219 pounds will receive a diet prescription of 1500 calories and 33 fat grams per day. Subjects weighing between 220 and 249 pounds will receive a diet prescription of 1800 calories and 40 fat grams per day. Subjects weighing greater than 250 pounds will receive a diet prescription of 2100 calories and 47 fat grams per day.
  Arms: Diet Only
Behavioral: Diet Plus Aerobic Training — Participants will receive all of the components as described for the DIET group. Additionally, this group will participate in supervised progressive aerobic training 3 days per week. Participants will be required to attend 3 sessions per week where they will participate in supervised exercise sessions progressing from 60 to 180 minutes per week of moderate-intensity (3.0-6.0 METS) aerobic exercise. 180 minutes per week of exercise will meet the American College of Sports Medicine and the American Heart Association recommendations of 450-750 METS.min.wk-1.
  Other Names: DIET+AT
  Arms: Diet plus Aerobic Training
Behavioral: Diet plus Resistance Training — Participants will receive all of the components as the DIET group. Participants will also participate in supervised resistance training protocol 3 days per week in the form of an individual session. The protocol will start the participants at a low volume of exercise at an intensity of 50-55% of 1-repetition maximum, and oscillate in both volume and intensity during the intervention, with a general trend toward increases in intensity as outlined in the ACSM Position Stand.
  Other Names: DIET+RT
  Arms: Diet plus Resistance Training

SUMMARY:
The purpose of this study is to examine the effect of weight loss and exercise on cardiovascular disease risk factors, specifically inflammation as measured by C-Reactive Protein and cardiac structure and function as measured by cardiac MRI, in Class II and III obese women during a 12 week training intervention.

DETAILED DESCRIPTION:
To date, research investigating obesity, inflammation, and cardiovascular disease has utilized lifestyle interventions focused on weight loss and exercise among groups with BMI classifications of normal, overweight and mildly obese. A limitation of recent investigations is the failure to utilize participants who are significantly overweight. Those whose BMI classification extends to Class II and Class III obesity (BMI > 35.0, and BMI > 40.0) have not yet been studied at length, yet these individuals have been shown to be able to substantially improve their cardiovascular risk profiles without attaining a BMI below 25. Inactivity has been linked to increased adiposity and a trend toward higher levels of cardiovascular disease risk. It is necessary to study the relationships between weight loss and weight loss with added physical activity among Class II and Class III obese participants in order to gain a more thorough knowledge of the effects of BMI on circulating markers of inflammation and the cardiac structural and functional changes associated with weight loss among this population. A second limitation of the current research is the use of strictly progressive resistance training protocols. The protocols used have increased constantly in intensity or volume, if not both. Constant increases in intensity tend to lead to overtraining among participants, highlighting a need for more variation of intensity and volume in the training protocol in order to avoid stagnation and overtraining. Finally, no research has studied the specific impact of diet and resistance training on either CRP or cardiovascular adaptations.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 30-55 years of age
* BMI = 35.0-44.9 kg/m2

Exclusion Criteria:

* Currently pregnant, pregnant in the past 6 months, or planning on becoming pregnant in the next 6 months.
* Regularly exercising for greater than 60 minutes per week.
* Taking prescription or over-the-counter medications that affect body weight, metabolism, blood pressure, or heart rate, such as psychotropic medications (e.g. zoloft, prozac, paxil, xanax) and medications that have metabolic effects (e.g. synthroid, wellbutrin, metformin).
* Having physical limitations that hinder or prevent exercise.
* Currently being treated for coronary heart disease, diabetes mellitus, hypertension, or cancer.
* Having a resting systolic blood pressure of > 150mmHg of diastolic blood pressure of > 100mmHg or currently taking any medications that affect blood pressure or heart rate (i.e. beta blockers).
* Currently enrolled in an exercise or weight control study or participating in an exercise or weight control study in the past 6 months.
* Have lost and not regained > 5% body weight in the past 6 months.
* Currently being treated for any psychological problems or taking any psychotropic medications.
* Abnormal kidney functions, as per current institutional standard for gadolinium administration.
* Known allergy to IV gadolinium, or the discovery of an allergic reaction to IV gadolinium at baseline.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Disease Risk Factors | 0 and 12 weeks
  Inflammation as determined by C-Reactive Protein and Cardiac Structure and Function as defined by left ventricular mass, aortic pulse wave velocity, fibrosis, and ejection fraction.

SECONDARY OUTCOMES:
Weight Loss | 0 and 12 weeks
  Weight loss by diet alone, diet plus aerobic training, and diet plus resistance training.

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Verba, MS, Principal Investigator — University of Pittsburgh; Blake D Justice, MS, Study Director — University of Pittsburgh
Locations (1):
- Physical Activity and Weight Management Research Center, Suite 600 Birmingham Towers, Pittsburgh, Pennsylvania, United States